CLINICAL TRIAL: NCT03249922
Title: A Prospective Analysis of Quality of Life Outcomes in Spinal Cord Stimulation
Brief Title: Quality of Life Outcomes in Spinal Cord Stimulation
Status: Terminated | Type: Observational
Why Stopped: Inadequate enrollment
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Antonios Mammis MD, Director, Center for Neuromodulation, Rutgers, The State University of New Jersey
Other Study IDs: Pro20170000766
Record Dates: First submitted 2017-08-11; First posted 2017-08-15 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Neuropathic Pain; Low Back Pain
Keywords: spinal cord stimulation
MeSH Terms: conditions — Neuralgia; Low Back Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Treatment Group: All patients who are considered candidates for spinal cord stimulator implant will be assigned to the "Treatment Group". Participiants will be clinically evaluated and given the Owenstry low back disability index, WHODAS 12, Beck depression index and SF-36.
  Interventions: Device: Spinal Cord Stimulation

INTERVENTIONS:
Device: Spinal Cord Stimulation — Implantation of a spinal cord stimulator for the control of axial back or neuropathic pain.

SUMMARY:
The investigators will be evaluating quality of life outcomes in patients who are undergoing routine spinal cord stimulator implant for uncontrolled pain. Patients will be evaluated pre and post-operatively for quality of life improvements, pain control, and functionality.

DETAILED DESCRIPTION:
This is a prospective cohort study for patients who will be undergoing implantation of spinal cord stimulator for pain. All patient will have implantation done at University Hospital Newark or Newark Beth Israel. The data points that will be collected will be the patient's weight, BMI, and detailed questionnaires regarding disability, activity, quality of life, and depression. The first data set will be taken pre-operatively at the DOC, 90 Bergen Street, suite 8100. Those patients enrolled will have the same data taken again upon subsequent postoperative visits at 3, 6, and 12 months. Being that spinal cord stimulation is a well-documented safe procedure, the investigators do not anticipate any deviation from the standard risks of surgery. With that being said the primary safety endpoint would be if there is an increased complication rate, secondary to the procedure, greater than the current anticipated risk rate. This is a purely observational study. Patients are not being recruited for an intervention but are being recruited during routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with neuropathic pain or axial back pain that is not controlled by oral analgesics, opioids, and has failed conservative management.
* Ages 18-90 with no ethnicity or gender predilections.

Exclusion Criteria:

* Patients who have spinal cord injury, multiple stimulator revisions, DRG stimulators, intrathecal pain pumps, complex regional pain syndrome, previous spinal cord stimulator implant, mechanical instability requiring fusion, myelopathy, psychological condition precluding them from complying with therapy, illegal drug abuse including heroin, cocaine, and illegally obtained prescription pills, or have previously been or are currently involved in litigation for medical malpractice.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients of the functional neurosurgery and neuromodulation department at New Jersey Medical School who present for indicated spinal cord stimulation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2018-07-22 (Actual); Study Completion 2018-07-22 (Actual)

PRIMARY OUTCOMES:
The number of patients with at least 50% improvement in VAS Pain Score | 12 Months
  The number of patients who had at least 50% improvement in VAS pain score
The number of patients with at least 50% improvement in Owenstry low back disability index | 12 Months
  The number of patients who had at least 50% improvement in disability as determined by this questionnaire.
The number of patients with at least 50% improvement in WHODAS 12 disability index. | 12 Months
  The number of patients who had at least 50% improvement in disability as determined by this questionnaire.

SECONDARY OUTCOMES:
The number of patients with at least 50% improvement in SF-36 quality of life score | 12 months
  The number of patients who had at least 50% improvement in quality of life as determined by this questionnaire.
The number of patients with at least 50% improvement in beck depression inventory | 12 Months
  The number of patients who had at least 50% improvement in depression as determined by this questionnaire.

OTHER OUTCOMES:
The Total number of surgical and post-operative Complications | 12 months
  Total number of surgical and post-operative complications occurring during the study

CONTACTS AND LOCATIONS:
Overall Officials: Antonios Mammis, MD, Principal Investigator — mammisan@njms.rutgers.edu
Locations (1):
- Neurologic Institute of New Jersey, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers.